CLINICAL TRIAL: NCT00867230
Title: A Phase I Open-Label Study of S-Trans, Trans-Farnesylthiosalicylic Acid (FTS) Administered on Days 1 to 21 of a 28 Day Cycle in Patients With Advanced Hematologic Malignancies
Brief Title: FTS Study in Patients With Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Concordia Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0201
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Myelodysplastic Syndrome; Leukemia
Keywords: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Agnogenic Myeloid Metaplasia; FTS; S-Trans, Trans-Farnesylthiosalicylic Acid
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis | interventions — farnesylthiosalicylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FTS (S-trans, trans-farnesylthiosalicylic acid) (Experimental)
  Interventions: Drug: FTS

INTERVENTIONS:
Drug: FTS — Starting dose of 100 mg twice a day by mouth, Days 1 through 21 of a 28-day cycle.
  Other Names: S-trans, trans-farnesylthiosalicylic

SUMMARY:
Primary Objective:

Determining the maximum tolerated dose (MTD) and pharmacokinetics (PK) of FTS (S-Trans, Trans-Farnesylthiosalicylic Acid) after daily oral administration on Days 1 through 21 of a 28-Day cycle to patients with advanced hematologic malignancies that have progressed following effective therapy or for which no effective therapy exists.

DETAILED DESCRIPTION:
FTS is designed to interfere with a cancer cell's ability to reproduce.

Before you can start receiving the drug on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your complete medical history will be recorded, and you will have a physical exam. You will be asked about any side effects that you are having and about any medications that you are taking. Your weight and vital signs (blood pressure, heart rate, breathing rate, and temperature) will be measured. Blood (about 2 tablespoons) and urine will be collected for routine tests. You will be asked about your ability to perform everyday tasks. You will have an electrocardiogram (ECG - test to measure the electrical activity of the heart). A bone marrow aspirate and/or biopsy will be collected to check the status of the disease. To collect a bone marrow aspirate and/or biopsy, an area of the hip or chest bone is numbed with anesthetic and a small amount (about 1 teaspoon) of bone marrow and bone is withdrawn through a large needle. Women who are able to have children must have a negative blood (about 1 tablespoon) or urine pregnancy test.

If you are found to be eligible for this study, you will take FTS by mouth, morning and night with food, on Days 1-21 of a 28-day study "cycle."

The amount of study drug you will receive will be based on when you enter the study. At least 3 participants will be taking FTS at the same dose level. Doses will be increased for the next group of 3 participants based on the side effects seen in the previous group. Each new group of participants will receive a higher dose level than the previous group, until a level is reached where side effects are considered to be intolerable.

After each cycle, your doctor may decide to increase your dose if you are not having intolerable side effects and you are benefitting from the study drug. If you experience intolerable side effects during any of the cycles of therapy with FTS, your dose may be reduced, delayed, or you may be taken off the study.

On Day 1 of the study, your weight and vital signs will be measured. Blood (about 1 tablespoon) will be collected for routine tests. You will not take your evening dose of FTS on Day 1.

On Days 8,15, and 22 of the first cycle, your weight and vital signs will be measured. You will be asked about any side effects that you are having, and about any medications that you are taking. On Day 15 of Cycle 1, blood (about 1 tablespoon) will also be drawn for routine tests.

During Cycle 1, on Days 1, 8, and 15, blood (about 1 tablespoon per draw) will be drawn to find out how much drug there is in your blood at different time points. This will help researchers to learn how FTS is processed by your body. This is called pharmacokinetic (PK) testing. Blood will be drawn before your morning dose of FTS, at 30, 60, and 90 minutes after taking the morning dose, and at 2, 4, 6, 8 and 24 hours after taking the morning dose. During Cycle 1, on Days 1 and 15, blood (about 3 tablespoons per draw) will be drawn to determine how FTS works against leukemia cells. This blood will be drawn before and 24 hours, after taking the morning dose on Day 1 and before you take the dose on Day 15.

On Day 1 of each cycle after Cycle 1, your weight and vital signs will be measured. Blood (about 2 tablespoons) and urine will be collected for routine tests. You will be asked about your ability to perform everyday tasks. You will be asked about any side effects that you are having, and about any medications that you are taking.

On Days 8, 15, and 22 of every cycle after Cycle 1, you will be asked about any side effects that you are having and about any medications that you are taking. On Day 15, blood (about 1 tablespoon) will also be drawn for routine tests, and your weight and vital signs will be measured.

You may remain on study for as long as you are benefiting. You will be taken off study if you are not benefitting or if you are experiencing intolerable side effects.

Thirty (30) days after you are no longer taking the study drug, you will have an end-of-study visit. Blood (about 2 tablespoons) and urine will be collected for routine tests. Your weight and vital signs will be measured. You will be asked about your ability to perform everyday tasks. You will be asked about any side effects that you are having, and about any medications that you are taking. You will have an ECG and an evaluation of your disease, which may include a bone marrow aspiration and/or biopsy.

This is an investigational study. FTS is not FDA approved or commercially available, and it has been authorized for use in research only. Up to 30 patients will take part in this multicenter study. Up to 20 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have relapsed/refractory hematologic malignancies for which no standard therapies are anticipated to result in a durable response or who have failed potentially curative therapy, or who refuse or are considered unsuitable for standard therapy. Patients with poor-risk myelodysplastic syndromes (MDS) [IPSS ≥ 1.5], chronic myelomonocytic leukemia (CMML), relapsed/refractory leukemias including
2. CONTINUATION OF # 1: acute myeloid leukemia (AML), acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), or chronic myelogenous leukemia (CML) in blastic phase, or with agnogenic myeloid metaplasia (AMM) are eligible.
3. Patients are eligible if they are 18 years or older
4. In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents, or at least 5 half-lives for noncytotoxic agents. If the patient is on hydroxyurea to control peripheral blood leukemic cell counts, the patient must be off hydroxyurea for at least 24 hours before initiation of treatment on this protocol. Persistent chronic clinically significant toxicities from prior chemotherapy must not be greater than Grade 1
5. Patients with active CNS disease are included and will be treated concurrently with intrathecal therapy
6. Patients must have ECOG performance status (PS) of 0 - 2
7. Have serum creatinine less than or equal to 2.0 mg/dl; total bilirubin less than or equal to 2.0 mg/dl; ALT and/or AST no more than 3X the upper limit of normal range unless abnormal parameter level is considered related to leukemia.
8. Patients must be willing and able to sign written informed consent and be able to comply with the study protocol for the duration of the study
9. Females of childbearing potential and males are required to practice adequate contraception or abstinence prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

1. Impaired cardiac function, including any one of the following: myocardial infarction within the previous 3 months; symptomatic coronary insufficiency or heart block; uncontrolled congestive heart failure; moderate or severe pulmonary dysfunction
2. Have an active uncontrolled infectious process
3. Significant impairment of gastrointestinal (GI) function of GI disease that may significantly alter the absorption of FTS(e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
4. Have received prior radiotherapy administered to more than 30% of marrow-bearing bone mass
5. Women patients are pregnant or lactating
6. Patients who have had major surgery without full recovery or major surgery within three weeks of FTS treatment start
7. Patients with marked baseline prolongation of QT/QTc interval (QTc interval greater than 480) using the Fridericia method as a main method of QTC analysis
8. Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Continous assessment throughout study and determination of dose limiting toxicities with each 28 day cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Laheru D, Shah P, Rajeshkumar NV, McAllister F, Taylor G, Goldsweig H, Le DT, Donehower R, Jimeno A, Linden S, Zhao M, Song D, Rudek MA, Hidalgo M. Integrated preclinical and clinical development of S-trans, trans-Farnesylthiosalicylic Acid (FTS, Salirasib) in pancreatic cancer. Invest New Drugs. 2012 Dec;30(6):2391-9. doi: 10.1007/s10637-012-9818-6. Epub 2012 May 1. PMID 22547163
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org